CLINICAL TRIAL: NCT05263336
Title: The Efficacy of Intraoperative ICG Angiography in Assuring Optimal Blood Supply to the Anastomosis in Rectal Cancer Patients Undergoing Laparoscopic Anterior Resection
Brief Title: Intraoperative Angiography Using ICG in Rectal Cancer Patients to Prevent Anastamotic Leak After Laparoscopic Anterior Resection of the Rectum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Paweł Bogacki, Principle Investigator, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICG UJ Krakow
Record Dates: First submitted 2022-01-27; First posted 2022-03-02 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; laparoscopic anterior resection; intraoperative angiography; ICG
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Intraoperative verdye green iv administration to visualize blood supply to the anastomosis
  Interventions: Drug: Verdye Green
- Control (No Intervention): No administration of verdye green intraoperatively

INTERVENTIONS:
Drug: Verdye Green — intraoperative iv application of indocyanic green for visualisation of blood supply to the anastomosis after rectal cancer recection
  Other Names: Indocyianic Green
  Arms: Intervention

SUMMARY:
The study enrols patients with operative rectal cancer qualified for laparoscopic anterior resection. Patients are given first dose of indocyanine green iv intraoperatively (ICG) before choosing the appropriate site of the anastomosis, and the second dose after performing the anastomosis to confirm adequate blood supply to the anastomotis. The main outcome assessed is the frequency o anastomotic leak in comparison to the group of patients that do not undergo intraoperative ICG angiography.

ELIGIBILITY:
Inclusion Criteria:

* operative rectal cancer

Exclusion Criteria:

* known allergy toward indocyanic green

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01-03 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Anastomotic leak | Up to two weeks post surgery
  Leakage in the anastomotic line defined as peritonitis requiring relaparotomy resulting from stool leakage from the anastomosis line

SECONDARY OUTCOMES:
Postsurgical Ileus | Up to 10 days post surgery
  Prolonged postsurgical ileus defined as no oral diet toleration, nausea, vomiting, no gas or stool passage lasting more than 4 days post surgery

CONTACTS AND LOCATIONS:
Locations (1):
- St John Grande Hospital, Krakow, Lesser Poland Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No